CLINICAL TRIAL: NCT02052167
Title: Human Factors Study for the Evaluation of the Methotrexate Prefilled Pen (50 mg/mL) for Subcutaneous Injection in Pediatric and Adolescent Patients With Juvenile Idiopathic Arthritis
Brief Title: Human Factors Study of Methotrexate Prefilled Pen (50 mg/mL) in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MC-MTX.16/HF Children
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate (Experimental)
  Interventions: Device: methotrexate prefilled pen

INTERVENTIONS:
Device: methotrexate prefilled pen

SUMMARY:
This study is planned to evaluate the human factor (HF)/usability of pediatric or adolescent JIA patients and the caregivers of Juvenile Idiopathic Arthritis (JIA) patients with the Methotrexate Prefilled Pen (including a label comprehension assessment and a device robustness evaluation).

ELIGIBILITY:
Main Inclusion Criteria:

* patient of either gender aged ≥2 to <21 years of age
* is a suitable candidate for treatment with injectable methotrexate for JIA per the patient's primary rheumatologist, with the previous or current diagnosis of active polyarticular course JIA

Main Exclusion Criteria:

* Is a female patient who is pregnant, trying to become pregnant, or breastfeeding, or of childbearing potential, sexually active but not practicing a highly reliable method of birth control during the study and at least 6 months thereafter
* Has contraindications for methotrexate
* Has a history of or current inflammatory arthritis or rheumatic autoimmune disease other than JIA
* Is unable, or does not have a caregiver able to comprehend written labeling and training materials

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of test case scenarios with observation and performance measures | 8 days
  Test case scenarios were designed to determine if the potential risks associated with the use of the prefilled pen were mitigated by information contained in the patient leaflet and the training provided to each patient or caregiver. The test case scenarios with observation and performance measures will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital & Clinics, Kansas City, Missouri, United States